CLINICAL TRIAL: NCT02871440
Title: A Two Comparator, Controlled Phase 3 Study of OM3 Tear Formulation Versus OPTIVE ADVANCED Unit Dose and OPTIVE Unit Dose Eye Drops in Patients With and Without Evaporative Dry Eye.
Brief Title: A Two Comparator, Controlled Phase 3 Study in Patients With and Without Evaporative Dry Eye
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of New South Wales (Other)
Collaborators: Allergan (Industry)
Responsible Party: Principal Investigator, Jacqueline Tan-Showyin, Research Fellow, The University of New South Wales
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOVS2016-040
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Results first posted 2020-05-12 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Dry Eye Syndromes
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Eye drop 1 (Experimental): Omega 3
  Interventions: Drug: Omega 3
- Eye drop 2 (Active Comparator): Optive Advanced
  Interventions: Drug: Optive Advanced
- Eye drop 3 (Active Comparator): Optive
  Interventions: Drug: Optive

INTERVENTIONS:
Drug: Omega 3
  Arms: Eye drop 1
Drug: Optive Advanced
  Arms: Eye drop 2
Drug: Optive
  Arms: Eye drop 3

SUMMARY:
Omega 3 (OM3) Tear is a new unit dose emulsion, containing flaxseed/castor oil, which is being developed by Allergan. It is desirable to understand the effect that this new emulsion has on tear film evaporation and tear lipid profile via interferometry, in patients with evaporative dry eye (EDE) and those without (non-EDE). It would also be valuable to evaluate the retention time of the lipid components of the new emulsion via tear collection and analysis in EDE and non-EDE patients

ELIGIBILITY:
Inclusion Criteria:

* Able to read and comprehend English and give informed consent as demonstrated by signing a record of informed consent;
* Over 18 years of age;
* Not wearing contact lenses in the past 3 months before enrolling
* Willing to use eye drops and comply with the study visit schedule as directed by the Investigator;
* Habitual (corrected or uncorrected) visual acuity of 6/9.5 or better in each eye;
* At the Screening visit (Day -14), patients must have Ocular Surface Disease Index (OSDI) score >18 (0 to 100 scale). At Baseline (Day 1) visits, patients must have OSDI score > 12 to continue in the study.
* TBUT≤10sec in at least 1 eye at Screening visit and Baseline visit
* Corneal sodium fluorescein staining score ≥ 1 and <4 (Oxford scheme) at Screening and Baseline visit.

Exclusion Criteria:

* Schirmer test (with anesthesia) ≤ 2 mm in either eye at Screening
* Patients who are currently using topical ocular medication or have used topical ocular medication within 2 weeks of the Screening visit. Patients who are being treated bilaterally with a marketed artificial tear for dry eye can be considered, provided they discontinue use at the Screening visit;
* Any active anterior segment disease excluding blepharitis;
* Any systemic disease that may affect ocular health e.g. Graves disease, and auto-immune diseases such as ankylosing spondylitis, multiple sclerosis and systemic lupus erythematosus;
* History of epilepsy or migraines exacerbated by flashing, strobe-like lights;
* Rigid or soft contact lens wearer, including orthokeratology;
* History of eye surgery within 6 months prior to enrolment in the study;
* Previous corneal refractive surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Stapleton, PhD, Study Director — University of New South Wales

RESULTS

PARTICIPANT FLOW:
Groups:
- Eye Drop 1: Omega 3 Tear Formulation (1-2 drops in each eye for at least 2 times daily)
- Eye Drop 2: Optive Advanced (1-2 drops in each eye for at least 2 times daily)
- Eye Drop 3: Optive (1-2 drops in each eye for at least 2 times daily)
Period: Overall Study
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3
Started | 12 | 13 | 15
Completed | 12 | 13 | 15
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3 | Total
Number analyzed (Participants) | 12 | 13 | 15 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 | 0 | 2
  Between 18 and 65 years | 10 | 8 | 10 | 28
  >=65 years | 1 | 4 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.98 (20.07) | 40.26 (20.84) | 40.91 (20.69) | 40.49 (20.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 11 | 9 | 26
  Male | 6 | 2 | 6 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 13 | 15 | 39
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 8 | 10 | 6 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 2 | 3 | 9 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 12 | 13 | 15 | 40
Ocular Surface Disease Index [Mean (Standard Deviation); unit: units on a scale] — Ocular Surface Disease Index has a score range of 0 to 100. Lower values indicate better outcomes.
  units on a scale | 35.28 (16.26) | 34.00 (14.34) | 34.47 (15.67) | 35.28 (16.14)
Tear Evaporation [Mean (Standard Deviation); unit: g/m^2*h] | 78.3 (42.8) | 67 (31.7) | 75.3 (38.0) | 78.0 (43.6)
Tear Break-Up Time [Mean (Standard Deviation); unit: seconds] | 6.14 (2.73) | 6.52 (2.95) | 6.22 (2.74) | 6.14 (2.73)
Tear Volume [Mean (Standard Deviation); unit: mm] — Schirmer's test is used to evaluate tear volume or tear production. Sterile paper strips are applied into the inferior-temporal aspect of the conjunctival sac of both eyes. The wetted length in millimeters is measures after 5 minutes.
  mm | 13.20 (9.06) | 13.83 (8.56) | 13.48 (8.93) | 13.83 (9.06)

OUTCOME MEASURES:

1. Primary Outcome: Tear Evaporation Rate
Description: Measured using a Vapometer (g/m^2*h)
Time Frame: Assessed at 4 weeks
Measure: Mean (Standard Deviation); unit: g/m^2*h
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3
Number analyzed (Participants) | 12 | 13 | 15
g/m^2*h | 77.7 (42.4) | 67 (31.7) | 75.3 (38.0)

2. Secondary Outcome: Tear Break-up Time
Description: Measured with fluorescein dye (seconds)
Time Frame: Assessed at 4 weeks
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3
Number analyzed (Participants) | 12 | 13 | 15
Seconds | 6.10 (2.76) | 6.52 (2.94) | 6.22 (2.73)

3. Secondary Outcome: Subjective Ocular Comfort
Description: Measured using visual analogue scales (0-100); 0 indicates no/less symptoms and 100 indicates maximum/worse symptoms.
Time Frame: Assessed at 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3
Number analyzed (Participants) | 12 | 13 | 15
score on a scale | 21 (23.73) | 21 (23.89) | 21 (23.73)

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: All-cause mortality or serious adverse events were monitored/assessed. Since, total number of participants at risk will equal the number of participants started in the participant flow module, this section has been updated.
Arm/Group | Eye Drop 1 | Eye Drop 2 | Eye Drop 3
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 3/12 | 4/13 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eye Drop 1 (N=12) | Eye Drop 2 (N=13) | Eye Drop 3 (N=15)
Bacterial Chest Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Itchy and uncomfortable eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Burning and Stinging in the eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Anemia and Vitamin D Deficiency (General disorders) | 1 (1) | 0 (0) | 0 (0)
Ocular irritation (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
Lid Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Dry white residue around the eyes 5 min after using study drops (Eye disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/40/NCT02871440/Prot_SAP_000.pdf